CLINICAL TRIAL: NCT02133872
Title: Angiotensin and Neuroimmune Activation in Hypertension
Brief Title: Study 1: Effect of Minocycline Treatment on Drug-Resistant Hypertensive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB2015005 -N; RO1HL3361028 (Other: NHLBI); 2013-00102 Study 1 (Other: UF IRB ID); 1R01HL132448-01 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
Keywords: Resistent Hypertension
MeSH Terms: conditions — Hypertension | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Open label, dose effectiveness trial
Oversight: Data Monitoring Committee: No

ARMS (3):
- Minocycline (50 mg/d) (Experimental): Subjects received minocycline 50mg/d.
  Interventions: Drug: Minocycline 50mg/d
- Minocycline (100 mg/d) (Experimental): Subjects received minocycline 50mg escalating to 100 mg/d.
  Interventions: Drug: Minocycline 100mg/d
- Minocycline (200 mg/d) (Experimental): Subjects received minocycline 50mg escalating to 100 mg then 200 mg/d.
  Interventions: Device: Minocycline 200mg/d

INTERVENTIONS:
Drug: Minocycline 50mg/d — Subjects will receive minocycline 50mg if no mean daytime ABPM SBP decline =/> 5mm Hg; subjects will receive minocycline 100mg, if no mean daytime ABPM SBP decline =/> 5mm Hg BP subjects will receive minocycline 200 mg.
  Arms: Minocycline (50 mg/d)
Drug: Minocycline 100mg/d — Subjects will receive minocycline 50mg if no mean daytime ABPM SBP decline =/> 5mm Hg; subjects will receive minocycline 100mg, if no mean daytime ABPM SBP decline =/> 5mm Hg BP subjects will receive minocycline 200 mg.
  Arms: Minocycline (100 mg/d)
Device: Minocycline 200mg/d — Subjects will receive minocycline 50mg if no mean daytime ABPM SBP decline =/> 5mm Hg; subjects will receive minocycline 100mg, if no mean daytime ABPM SBP decline =/> 5mm Hg BP subjects will receive minocycline 200 mg.
  Arms: Minocycline (200 mg/d)

SUMMARY:
Hypertension (HTN) is the single most prevalent risk factor for cardiovascular disease, diabetes, obesity and metabolic syndrome. Recent American Heart Association (AHA) statistics indicate that one-third of all adults in the United States of America suffer from HTN. Despite advances in life style modification and multi-drug therapies, 20-30% of all hypertensive patients remain resistant.

These individuals exhibit autonomic dysregulation due to elevated sympathetic activity and norepinephrine spillover, and low parasympathetic activity. It is generally accepted that this uncontrolled, resistant HTN is primarily "neurogenic" in origin, involving over activity of the sympathetic nervous system that initiates and sustains HTN. A surgical approach such as the recently developed "Simplicity Catheter" assisted renal denervation remains one of the few options available to these patients. Thus, a mechanism-based breakthrough is imperative to develop novel strategies to prevent and perhaps eventually cure neurogenic hypertension (NH). This study is designed to evaluate a low and high dose of minocycline to test the hypothesis that minocycline treatment would produce antihypertensive effects in drug-resistant neurogenic hypertensive individuals. Minocycline has been selected because of its demonstrated effects on inhibiting microglial activation and its ability to penetrate the blood brain barrier. There is no other compound available that is safer and displays specificity better than Minocycline in inhibiting microglial activation. Thus, the potential therapeutic benefits of this inexpensive, well tolerated, already FDA-approved drug that has minimal side effects would be enormous.

DETAILED DESCRIPTION:
Open-label design of dose titration for each participant beginning at 50 mg/day of minocycline, escalating to 100 mg/day and 200 mg/day if the primary outcome measure of ambulatory blood pressure monitor (ABPM) =/> to 5 mmHg decrease in mean daytime SBP was not achieved. If patients responded, participation was completed. This revised protocol was resubmitted to the IRB and approved on 1/6/16. An interim analysis was planned after 40 patients completed the revised protocol.

In addition to blood collection, a physical exam will be conducted and office systolic blood pressure (BP), diastolic blood pressure (DBP) and pulse pressure (PP) will be recorded. Patients will be fitted with an ABPM system. Patients will wear the ABPM for 24 hours at which point they will mail the monitor back to research personnel. At this visit, the study drug will be dispensed and patients will be instructed to start the study medication after completing the 24- hour ABPM monitoring period. After this visit, patients will be asked to return every month till the end of the study at 6 months.

Monthly visits (1, 2, 3, 4, 5 and 6 month visits), will include a brief physical examination and an assessment of medication compliance and tolerance. One tablespoon of blood will be drawn for flow cytometry analysis, selected cytokines, markers of gut permeability including zonulin, and iPSCs isolation at the baseline, 3 and 6 month visit only. Study drug will be dispensed and measurement of SBP, DBP, PP and other vital signs will also be completed. Office BP readings will be taken in a seated position after 5 minutes of rest according to Joint National Committee VII Guidelines. At baseline, BP will be measured at each arm, and the arm with the higher BP will be used for all subsequent readings. Averages of the triplicate measures will be calculated and used for analysis. At baseline and each followup visit, patients will be asked to wear the ABPM for 24 hours. Subjects will mail the cuff back to research personnel when completed. ABPM will be performed using an oscillometric Spacelabs 90207 monitor (Spacelabs Healthcare, Issaqua, WA) with readings taken every 30 minutes in daytime and every 60 minutes at nighttime. ABPM readings will be averaged for, daytime and nighttime. Patients will be assessed while adhering to their usual diurnal activity and nocturnal sleep routine. The antihypertensive drugs, and their doses, used at each visit will be recorded on standardized forms along with any reports of adverse experiences known to occur with the drugs used (e.g. lightheadedness, dizziness, syncope, etc.).

If patients respond to treatment, by protocol defined drop in daytime ABPM and/or the need for down titration of hypertensive therapy they will be considered a responder, complete the final visit and complete study participation. At the final visit, the same blood tests at baseline will be repeated. When the patients complete the 6 months of treatment or are considered a responder at a lower dose, they will come in for their final visit, and return the ABPM monitor, their participation in the trial will be considered as complete.

ELIGIBILITY:
Inclusion:

* Greater than 18 and less than 86 years of age;
* On stable medication regimen
* Full-tolerated doses of 3 or more antihypertensive medications of different classes, one of which must be a diuretic (with no changes for a minimum of two months prior to screening) that is expected to be maintained without changes for at least 3 months.
* The individual agrees to have all study procedures performed
* Willing to provide written consent

Exclusion

* eGFR of < 45mL/min/1.73m2, using the MDRD calculation.
* More than one in-patient hospitalization for an antihypertensive crisis within the year.
* More than one episode(s) of orthostatic hypotension (reduction of SBP of ≥ 20mmHg of diastolic blood pressure (DBP) of ≥ 10mmHg within 3 minutes of standing).
* Known hypersensitivity or contraindication to Minocycline or other tetracycline.
* Evidence of alcoholism or drug abuse;

  * Concurrent severe disease (such as neoplasm or HIV positive or AIDS).
  * Women of childbearing potential

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cardiovascular Clinic, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label design of dose titration. Subjects will receive minocycline 50mg if no mean daytime ABPM SBP decline =/> 5mm Hg; subjects will receive minocycline 100mg, if no mean daytime ABPM SBP decline =/> 5mm Hg BP subjects will receive minocycline 200 mg.
Groups:
- Minocycline (100 mg/d): Subjects received minocycline 50mg escalated to 100 mg/d.
Period: Overall Study
Arm/Group | MInocycline (50 mg/d) | Minocycline (100 mg/d) | Minocycline (200 mg/d)
Started | 15 | 5 | 14
Completed | 10 | 2 | 14
Not Completed | 5 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The total population of subjects in the Minocycline Dose Escalation is 34. Arms/Groups are Combined to describe total population of 34 subjects. 34 subjects started study and only these 34 moved through study arms as follows: Non-Responders of 50 mg/d continued to 100 mg/d. Non-responders of 100 mg/d continued to 200 mg/d.
Groups:
- Minocycline Dose Escalation: The total population of subject in the Minocycline Dose Escalation is 34. Non-Responders of 50 mg/d continued to 100 mg/d. Non-responders of 100 mg/d continued to 200 mg/d.
Arm/Group | Minocycline Dose Escalation
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.06 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34
Baseline office SBP [Mean (Standard Deviation); unit: mmHg] | 140 (14)

OUTCOME MEASURES:

1. Primary Outcome: Categorical Classification of Subjects Into Responders vs. Non-responders
Description: The primary measure of interest was the categorical classification of subjects into responders vs. non-responders upon treatment with a specific minocycline dose: 50, 100 or 200 mg/d. Responders are defined as subjects who achieve a drop of >5 mmHg in mean daytime SBP, based on daytime ABPM measurements (7 am to 10 pm). For these participants, the discontinuation or lowering of the dose of a concurrent anti-hypertensive drug due to excessive SBP reduction will also be assessed. Excessive SBP reduction is defined as an office SBP <120 mmHg or >10 mmHg SBP decrease associated with symptom(s). On the other hand, non-responders are defined as the participants that fail to show any change in their average daytime SBP measured through ABPM despite being exposed to the different minocycline doses evaluated.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Minocycline (50 mg/d) | Minocycline (100 mg/d) | Minocycline (200 mg/d)
Number analyzed (Participants) | 34 | 19 | 14
Participants
  Responders | 10 | 2 | 4
  Non-responders | 19 | 14 | 10
  Participants who withdrew from study | 5 | 3 | 0

2. Secondary Outcome: Change in 24 Hour SBP by ABPM
Description: Among Responders, difference in overall daytime and nighttime Systolic Blood Pressure (SBP) using 24 hour Ambulatory Blood Pressure Monitoring (ABPM) from baseline to final visit
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Minocycline (50 mg/d) | Minocycline (100 mg/d) | Minocycline (200 mg/d)
Number analyzed (Participants) | 10 | 2 | 4
mmHg | 4 (12) | 4 (3) | 16 (3)

3. Secondary Outcome: Changes in Office SBP Over Time
Description: Among Responders, evaluation of changes in office systolic blood pressure (SBP) from baseline to final visit
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Minocycline (50mg/d): Subjects received minocycline 50mg/d.
Arm/Group | Minocycline (50mg/d) | Minocycline (100 mg/d) | Minocycline (200 mg/d)
Number analyzed (Participants) | 10 | 2 | 4
mmHg | 13 (10) | 2 (1) | 20 (16)

ADVERSE EVENTS:
Time Frame: 180 days - from baseline to final visit
Arm/Group | Minocycline (50 mg/d) | Minocycline (100 mg/d) | Minocycline (200 mg/d)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/5 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/5 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 2/5 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocycline (50 mg/d) (N=15) | Minocycline (100 mg/d) (N=5) | Minocycline (200 mg/d) (N=14)
Asymptomatic hypotension (Vascular disorders) | 3 (3) | 2 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02133872/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02133872/ICF_001.pdf